CLINICAL TRIAL: NCT05302492
Title: Feasibility of Improvement for Elderly Sleep Disturbance Through Home Care Solution
Brief Title: Elderly Sleep Disturbance Through Home Care Solution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202100552A3
Record Dates: First submitted 2022-02-11; First posted 2022-03-31 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2023-05

CONDITIONS: Aging; Sleep Disturbance
Keywords: aging; sleep disturbance; CPAP; phototherapy; omics
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep apnea group with CPAP (Experimental): Intervention group: CPAP for 3 months in elderly diagnosis with sleep apnea and AHI > 15/h.
  Control group: sleep apnea and patient refuse treatment or poor compliance.
  Interventions: Device: CPAP
- sleep disturbance without sleep apnea nor PLMS (Experimental): Intervention group: light box on elderly with sleep disturbance with PSQI > 5 and no OSA and no PLMS control group: elderly with sleep disturbance with PSQI > 5 and no OSA and no PLMS refuse light box or poor compliance
  Interventions: Device: Light box

INTERVENTIONS:
Device: CPAP — CPAP: continue positive airway pressure ventilator is the standard treatment of OSA.
  Arms: Sleep apnea group with CPAP
Device: Light box — Light box: is the treatment choice for circadian rhythm disorders. now apply to sleep disturbance without OSA or PLMS.
  Arms: sleep disturbance without sleep apnea nor PLMS

SUMMARY:
Humans spend a third of their time on sleep. Therefore, maintaining a deep, stable and consistent sleep is very important for a good quality of life. Aging is often related to a decrease in the ability to fall asleep and maintain sleep. Getting older, various factors can worsen the normal sleep process, which is essential for restoring function and body function. Aging-related diseases, life changes, or own aging can disrupt the normal sleep cycle and seriously affect healthy aging. For example, the circadian rhythm and sleep consolidation will be broken with normal aging. These changes may lead to aging, or become part of the risk factors for diseases such as Alzheimer's disease. How to avoid disability and dementia by improving the quality of sleep to make the elderly healthy and aging, will bring huge effects to the economy, society, and health care.

From this plan, investigators will participate in an integrated plan (main plan)-" Integrating Systematic Data of Geriatric Medicine to Explore the Solution for Healthy Aging". In the main plan, 500 subjects will be enrolled. All subjects consent to provide medical record and will be tested for sarcopenia, including body composition, 4-meter walk, handgrip strength. The subjects screened sleep-affected subjects. It is estimated that 250 people will be invited for home sleep testing, such as continuous positive pressure breathing aid (CPAP) for sleep apnea (OSA) (approximately 120 subjects). For non-OSA and non-periodic limb movement disorder (PLMS) sleep problems, take a phototherapy program (about 60 subjects). The following goals are expected to be achieved:

1. Link to the main project to explore the correlation between common sleep disorders in the elderly and blood pressure, cognition, sarcopenia, metabolomics or intestinal microbiome
2. To verify the prognosis of sleep apnea and sleep disorders after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Those who are willing to sign the written subject consent
* Participants who participated in the integrated project (main project) - "Integrating Systematic Data of Geriatric Medicine to Explore the Solution for Healthy Aging"
* The results of the sleep questionnaire meet one of the following:

  1. Pittsburgh Sleep Quality Scale (PSQI) > 5 points
  2. The Self-Sleep Assessment Questionnaire (STOP-BANG) is at high risk for sleep apnea (OSA)

Exclusion Criteria:

* Patients with severe cataracts who have not received treatment, patients with color blindness and chronic skin diseases (including psoriasis, eczema), or those who are considered by the host to be unable to receive light therapy.
* Those who are unsuitable after evaluation by a physician.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 107 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline PSQI ( Pittsburg Sleep Quality Index ) at 3 months | 3 months
  Subjective sleep quality will be assessed by the PSQI questionnaire. The measure consists of 19 individual items, creating 7 components that produce one global score. Each component is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.

SECONDARY OUTCOMES:
Change from baseline sleep efficiency at 3 months | 3 months
  The sleep efficiency, defined as the percent of time scored as sleep during the sleep period, was calculated as a daily average from one week of actigraphy recordings. Increased sleep efficiency will be identified as improved objective sleep quality.
Change from baseline total sleep time at 3 months | 3 months
  The total sleep time, defined as the minutes of sleep between sleep onset and wake time, was calculated as a daily average from one week of actigraphy recordings. Increased total sleep time will be identified as improved objective sleep quality.
Change from baseline sleep onset latency at 3 months | 3 months
  The sleep onset latency, defined as the minutes between lights off and first sleep episode, was calculated as a daily average from one week of actigraphy recordings. Decreased sleep onset latency will be identified as improved objective sleep quality.
Change from baseline wake after sleep onset (WASO) at 3 months | 3 months
  The WASO, defined as the minutes awake during the sleep period after sleep onset, was calculated as a daily average from one week of actigraphy recordings. Decreased WASO (wake after sleep onset) will be identified as improved objective sleep quality.
Change from baseline appendicular skeletal muscle mass at 3 months | 3 months
  The appendicular skeletal muscle mass was evaluated by body composition analysis.(Tanita MC-780 MA)
Change from baseline handgrip strength at 3 months | 3 months
  The handgrip strength (kg) was evaluated by Hand Dynamometer. (Jamar® Plus+ Digital Hand Dynamometer)
Change from baseline gait speed at 3 months | 3 months
  The gait speed test was performed by recording the average time of walking 4 meters and representing with the distance (m) per second.

CONTACTS AND LOCATIONS:
Overall Officials: Ning-hong Chen, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan